CLINICAL TRIAL: NCT00157573
Title: Phase II Trial of GM-CSF in Women With Asymptomatic Ovarian, Primary Peritoneal, or Tubal Carcinoma
Brief Title: GM-CSF, Sargramostim in Women With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Bayer (Industry)
Responsible Party: Principal Investigator, Richard Thomas Penson, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 04-305
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer
Keywords: Asymptomatic; Clinical trial; Phase II; GM-CSF; Immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GM-CSF, Sargramostim Cohort 1 (Experimental): GM-CSF, Sargramostim 250 μg/m^2 subcutaneous injection daily on days 1 to 14 in a 28-day cycle until disease progression or unacceptable toxicity for a median of 3 cycles.
  Interventions: Drug: GM-CSF, sargramostim
- GM-CSF, Sargramostim Cohort 2 (Experimental): GM-CSF, sargramostim 150 μg/m^2 subcutaneous injection daily for 28 days in a 28-day cycle until disease progression or unacceptable toxicity fora median of 3 cycles. GM-CSF, sargramostim dose escalation was permitted up to 250 μg/m^2 per day if applicable based on toxicity and white blood cell count.
  Interventions: Drug: GM-CSF, sargramostim

INTERVENTIONS:
Drug: GM-CSF, sargramostim — GM-CSF subcutaneous injection
  Other Names: Leukine®

SUMMARY:
Granulocyte macrophage colony-stimulating factor (GM-CSF) is an immunostimulant and preliminary data suggests it may change the natural history of prostate cancer and melanoma. This study looks at ability of GM-CSF to alter disease progression in women who have recurrent but asymptomatic recurrence of their ovarian cancer.

DETAILED DESCRIPTION:
This is an open labeled, single arm phase II study of GM-CSF, sargramostim delivered daily without a break in a population of healthy and fit women with evidence of recurrent but asymptomatic mullerian malignancy (such as ovarian cancer, fallopian tube cancer, or primary peritoneal cancer). The main goal is to determine the time to treatment termination due to disease progression or toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of histologic or cytologic diagnosis of primary ovarian, primary peritoneal or tubal carcinoma.
* Patients must be asymptomatic from their cancer.
* Patients must have evidence of recurrent carcinoma, as determined by:

  * A rising cancer antigen 125 (CA-125) serum level greater than 35 U/mL or two successive rising values with the most recent value at least 3 times the nadir value.
  * Or evidence of evaluable or measurable disease by x-ray or computed tomography (CT) scan.
* Patients may not receive concurrent antineoplastic therapy. All hormonal therapy used as a treatment modality (i.e. tamoxifen, arimidex, etc) must be stopped prior to treatment on protocol.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.

Exclusion Criteria:

* Known severe hypersensitivity to GM-CSF.
* Other coexisting malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma or cervical cancer in situ or concurrent superficial or stage IB endometrial carcinoma.
* Concomitant use of anti-neoplastic therapy.
* Treatment with a non-FDA approved or investigational drug within 30 days before Day 1 of trial treatment.
* Any unresolved chronic toxicity greater then Common Toxicity Criteria (CTC) grade 2 from previous anticancer therapy (except alopecia).
* Serum creatinine level greater than CTC grade 2 [1.5 x upper limit normal (ULN)].
* Pregnancy or breast feeding (women of childbearing potential).
* Severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) as judged by the investigator.
* Significant clinical disorder or laboratory finding that makes it potentially unsafe for the subject to participate in the trial as judged by the investigator.
* Patients currently receiving other investigational antineoplastic agents, on systemic chemotherapy or under radiation therapy treatment.
* Patients with clinical and/or radiographic evidence of current or impending bowel obstruction.
* Performance status < 1.
* Ability to understand and the willingness to sign a written informed consent document.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-12; Primary Completion 2008-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Penson, M.D., Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Result] Roche MR, Rudd PJ, Krasner CN, Matulonis UA, Berlin ST, Lee H, Silver M, Tran CD, Seiden MV, Penson RT. Phase II trial of GM-CSF in women with asymptomatic recurrent mullerian tumors. Gynecol Oncol. 2010 Feb;116(2):168-72. doi: 10.1016/j.ygyno.2009.10.075. Epub 2009 Nov 18. PMID 19922985
- See also: Sponsor information — http://www.dfhcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Granulocyte macrophage colony-stimulating factor (GM-CSF) Phase II recruitment from oncology clinic.
Pre-assignment Details: Phase II
Groups:
- GM-CSF, Sargramostim Cohort 2: GM-CSF, sargramostim 150 μg/m^2 subcutaneous injection daily for 28 days in a 28-day cycle until disease progression or unacceptable toxicity for a median of 3 cycles. GM-CSF, sargramostim dose escalation was permitted up to 250 μg/m^2 per day if applicable based on toxicity and the white blood cell count.
Period: Overall Study
Arm/Group | GM-CSF, Sargramostim Cohort 1 | GM-CSF, Sargramostim Cohort 2
Started | 35 | 37
Completed | 35 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 72 ovarian cancer patients with evaluable or measurable disease.
Groups:
- GM-CSF, Sargramostim: All enrolled eligible participants who participated in Cohort 1 or Cohort 2 of the study.
  In Cohort 1 participants received GM-CSF, sargramostim 250 μg/m^2 subcutaneous injection daily on days 1 to 14 in a 28-day cycle until disease progression or unacceptable toxicity for a median of 3 cycles.
  In Cohort 2 participants received GM-CSF, sargramostim 150 μg/m^2 subcutaneous injection daily for 28 days in a 28-day cycle until disease progression or unacceptable toxicity for a median of 3 cycles. GM-CSF, sargramostim dose escalation was permitted up to 250 μg/m^2 per day if applicable based on toxicity and white blood cell count.
Arm/Group | GM-CSF, Sargramostim
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Treatment Termination (TTT)
Description: TTT is the median time in days to discontinuing treatment with GM-CSF, sargramostim (treatment termination) e.g. time on study until progression of disease, unacceptable adverse effects, bowel obstruction, development of new ascites or pleural effusions, initiation of systemic chemotherapy, participant death, development of co-morbid diseases which make participant continuation on the trial unsafe in the judgment of the principal investigator or the treating physician or withdrawal of consent by the participant.
Time Frame: Up to 460 days
Population: After initial analysis, it was clear that the schedule did not significantly impact the immune response and that the actual white cell count (WCC) was the best correlate predictor of change in CA125, and so the cohorts were combined for an overall analysis. 1 participant withdrew consent and was not included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | GM-CSF, Sargramostim
Number analyzed (Participants) | 71
days | 78 [14 to 460]

2. Secondary Outcome: Median Time to Progression (TTP)
Description: TTP was defined as the median time in days from trial entry until progressive disease (PD) was documented as defined by RECIST criteria. PD was defined of at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In participants with no measurable disease who had an informative cancer antigen-125 (CA-125), PD was defined as a rise of > 50% over Baseline, confirmed by a subsequently higher value at least 21 days later.
Time Frame: Up to 60 months
Population: No analysis was performed. No data was reported for TTP in the clinical chart that was found to be reliable or consistent in the absence of proper computed tomography (CT) surveillance.
Arm/Group | GM-CSF, Sargramostim
Number analyzed (Participants) | 0

3. Secondary Outcome: Tumor Response Rate (RR)
Description: RR is the percentage of patients with response as assessed by the investigator using Response Evaluable Criteria in Solid Tumors (RECIST) and CA-125 Rustin criteria. Complete Response (CR) is the disappearance of all target and non-target lesions and normalization of CA-125. Partial Response (PR) is at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; in patients with no measurable disease with an informative CA-125, the 75% definitions by Rustin is used. Stable Disease is neither sufficient shrinkage for PR nor increase for PD, taking as reference the smallest sum LD since the treatment start. PD is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since treatment start or the appearance of one or more new lesions; in patients with no measurable disease with an informative CA-125, PD is defined as a rise of > 50% over baseline, confirmed by a higher value 21 days later.
Time Frame: Up to 60 months
Population: After initial analysis, it was clear that the schedule did not significantly impact the immune response and that the actual WCC was the best correlate predictor of change in CA125, and so the cohorts were combined for an overall analysis. 1 participant withdrew consent and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF, Sargramostim
Number analyzed (Participants) | 71
Participants
  Complete Response | 1
  Partial Response | 0
  Stable Disease | 20
  Progressive Disease | 50

4. Secondary Outcome: Number of Participants With Adverse Events (Toxicity) Grade 3 or 4
Description: Adverse Events (previously toxicity) were graded according the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 3.0. The total number of participants with adverse events graded 3 (severe) or 4 (life-threatening or disabling) are reported.
Time Frame: Up to 460 days
Population: After initial analysis, it was clear that the schedule did not significantly impact the immune response and that the WCC was the best correlate predictor of change in CA125, and so the cohorts were combined for an overall analysis. 1 participant withdrew consent and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF, Sargramostim
Number analyzed (Participants) | 72
Participants
  Thrombocytopenia | 2
  Musculoskeletal pain | 9
  Fatigue | 3
  Abnormal liver function test | 2
  Vomiting | 2
  Metabolic | 2
  Small bowel obstruction | 2
  Myelodysplasia | 1
  Urticaria | 1
  Abdominal pain | 1
  Palpitations | 1
  Hypertension | 1
  Changes in bowel habit | 1
  Diverticulitis | 1
  Gout | 1
  Headache | 1
  Macular tuft | 1
  Nausea sinus | 1
  Bradycardia | 1

5. Other Pre Specified Outcome: Change From Baseline of Anti-Trag Antibodies
Time Frame: Up to 60 months
Population: This outcome measure was originally posted as a secondary outcome measures but was actually an exploratory endpoint. No data was collected.
Arm/Group | GM-CSF, Sargramostim
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Between December 2004 and October 2008, 72 eligible and evaluable patients were enrolled. Adverse events (AEs) were collected for 30 calendar days after administration of the last dose of trial drug (Up to 234 days)
Groups:
- GM-CSF, Sargramostim Cohort 2: GM-CSF, sargramostim 150 μg/m^2 subcutaneous injection daily for 28 days in a 28-day cycle until disease progression or unacceptable toxicity for a median of 3 cycles. GM-CSF dose escalation was permitted up to 250 μg/m^2 per day if applicable based on toxicity and white blood cell count.
Arm/Group | GM-CSF, Sargramostim Cohort 1 | GM-CSF, Sargramostim Cohort 2
Serious Adverse Events (participants affected / at risk) | 2/35 | 5/37
Other Adverse Events (participants affected / at risk) | 35/35 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF, Sargramostim Cohort 1 (N=35) | GM-CSF, Sargramostim Cohort 2 (N=37)
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bowel obstruction (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF, Sargramostim Cohort 1 (N=35) | GM-CSF, Sargramostim Cohort 2 (N=37)
Allergic reaction (Skin and subcutaneous tissue disorders) | 35 | 36
Hemoglobin (Blood and lymphatic system disorders) | 2 | 0
Leukocytes (Blood and lymphatic system disorders) | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Fatigue (General disorders) | 35 | 19
Fever without neutropenia (General disorders) | 35 | 36
Rigors/Chills (General disorders) | 6 | 2
Weight loss (Investigations) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Injection site reaction (Skin and subcutaneous tissue disorders) | 26 | 28
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Hot flashes (Endocrine disorders) | 6 | 1
Anorexia (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 11 | 7
Dehydration (Gastrointestinal disorders) | 2 | 0
Diarrhea without prior colostomy (Gastrointestinal disorders) | 9 | 8
Esophagitis (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 9 | 10
Vomiting (Gastrointestinal disorders) | 9 | 3
Alkaline phosphatase (Investigations) | 2 | 1
Alanine aminotransferase (Investigations) | 3 | 2
Aspartate aminotransferase (Investigations) | 3 | 1
Hyperglycemia (Investigations) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 0
Abdomen pain (Gastrointestinal disorders) | 10 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 35 | 36
Chest wall pain (General disorders) | 5 | 1
Extremity limb pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Headache (Nervous system disorders) | 12 | 8
Joint pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary/upper respiratory other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Platelets (Blood and lymphatic system disorders) | 1 | 2
Hematologic-other (Blood and lymphatic system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 3
Distention/bloating abdominal (Gastrointestinal disorders) | 1 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gastrointestinal other (Gastrointestinal disorders) | 0 | 2
Sinus Infection (Infections and infestations) | 0 | 2
Edema limb (Metabolism and nutrition disorders) | 0 | 4
Neuropathy sensory (Nervous system disorders) | 1 | 13
Ocular other (Eye disorders) | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 3
Pain other (General disorders) | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Incontinence urinary (Renal and urinary disorders) | 0 | 2
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No